CLINICAL TRIAL: NCT02622542
Title: A Randomized Controlled Comparative Study on Effectiveness of Endovascular Repair Versus Best Medical Therapy for Acute Uncomplicated Type B Aortic Dissection
Brief Title: ACute Uncomplicated Type b Aortic Dissection: Endovascular Repair vs. Best Medical Therapy
Acronym: ACUTE-B
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Harleen K Sandhu, Associate Professor, Department of Cardiothoracic and Vascular Surgery, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTVS-KC03; HSC-MS-15-0937 (Other: University of Texas Health Science Center at Houston IRB)
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Distal Aortic Dissection; Dissection, Aortic Acute; Acute Type B Aortic Dissection (Uncomplicated)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participant and investigator/treating physician would be blinded until the day of treament initiation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BMT Alone (Active Comparator): Patients in this group will be managed with the best medical therapy (BMT) alone
  Interventions: Other: BMT
- BMT+TEVAR (Experimental): Patients in this group will be managed with thoracic endovascular aortic repair (TEVAR) in addition to the best medical therapy (BMT)
  Interventions: Device: BMT+TEVAR

INTERVENTIONS:
Device: BMT+TEVAR — These FDA-approved devices will be used for performing TEVAR in the patients randomized to this arm, in addition to the medical therapy to control blood pressure (BMT)
  Other Names: Medtronic® Valiant® Thoracic Stent Graft; Conformable GORE® TAG® Thoracic Endoprosthesis
  Arms: BMT+TEVAR
Other: BMT — Optimal medical therapy will be administered to the patients randomized to this arm, involving but not limited to, beta-blockers, etc., to control the blood pressure and pain for stabilizing the patient upon presentation.
  Arms: BMT Alone

SUMMARY:
The purpose of the study is to conduct a randomized controlled trial comparing best medical therapy (BMT) alone to BMT with thoracic endovascular aortic repair (BMT+TEVAR) for uncomplicated acute type B aortic dissection.

DETAILED DESCRIPTION:
Study Design:

This is a prospective, two-arm, parallel-group, single-center, pragmatic, randomized clinical trial.

Population:

The target population comprises all adult patients aged 18 years and older who present with uncomplicated acute type B aortic dissection. The study sample will include 436 subjects of both genders and any race or ethnicity.

Procedures:

Eligible and consented patients will be enrolled into the study if all eligibility criteria are met and will be randomly allocated to one of the two study arms: BMT vs BMT+TEVAR

Study Duration:

The study is expected to accrue patients over the course of 5 years and total follow up per patient for 5 years. Overall duration of the study is anticipated to be about 10 years for completion of all study endpoints.

Endpoints:

* Primary Outcome: To determine all-cause mortality among both study arms.
* Secondary Outcomes: To assess any major morbidity events (rupture, aortic intervention or reintervention, progression to complicated dissection, aneurysm formation, malperfusion resulting in organ failure, and aorta-specific mortality), as will quality of life measures, temporal discounting assessment and outcomes comparison in an observational cohort of patients who decline to be randomized due to a strong treatment preference.

Risks and Benefits:

Since this study involves only usual care and FDA-approved treatments, the investigators do not expect any additional physical risks to patients beyond those associated with usual care. One discernible risk involved in study participants is an unintentional disclosure of sensitive patient health information.

The participants of this study do not stand to benefit directly from taking part. However, the investigators hope that the results obtained from this study would provide useful information that would help delineate a standard and economical management protocol for acute Type B aortic dissection in future.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years, regardless of race or ethnicity;
* Diagnosed with uncomplicated ABAD, i.e., a primary entry tear distal to left subclavian artery with no evidence of malperfusion, end-organ ischemia, rupture, or intractable pain, and onset of symptoms is ≤30 days prior to enrollment;
* Patient has been stabilized after the acute event with control of pain and blood pressure using ≤3 intravenous antihypertensive medications;
* Adequate imaging, e.g., CT with contrast (chest + abdomen+ pelvis) is available prior to enrollment; and
* Indicates willingness to comply with the study protocol and is able to provide a written informed consent;
* Meets criteria for inclusion in the National Death Index and Social Security Death Master File.

Exclusion Criteria:

* Diagnosed with Type A aortic dissection;
* Evidence of complicated ABAD;
* Chronic Type B aortic dissection (>6 weeks from onset of symptoms);
* Unable to be randomized and undergo treatment according to protocol within 30 days of symptom onset;
* Diagnosed with traumatic dissection or penetrating ulcer;
* Anatomy is not suitable for TEVAR;
* Previous descending thoracic or abdominal aortic surgery (open or endovascular);
* Unsuitable access sites, including infection at access sites;
* Associated aortic aneurysm (descending aortic diameter ≥5.0 cm);
* Life expectancy <2 years;
* Unable or unlikely to comply with BMT;
* Unable or refuse to comply with follow-up;
* Intend to participate in another trial within 3 months of enrollment;
* Pregnant or breast-feeding;
* Vasculitis or known genetic connective tissue disorder (Marfan's syndrome or Ehlers-Danlos syndrome)
* Active systemic infection;
* Chronic kidney disease stage 3-5 (estimated glomerular filtration rate <60 mL/min/1.73m2);
* Cerebral vascular accident within past 3 months; or
* Clinically significant gastrointestinal bleeding, major surgery, myocardial infarction, or untreated coagulopathy within past 6 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 5 years
  Participants would be followed for a period of 5 years following initial presentation

SECONDARY OUTCOMES:
Any major morbidity events | 5 years
  Participants would be followed for a period of 5 years following initial presentation to record any major events (rupture, aortic intervention or reintervention, progression to complicated dissection, aneurysm formation, malperfusion resulting in organ failure, and aorta-specific mortality)
Change in Quality of Life assessment | 5 years
  Participants would be followed for a period of 5 years following initial presentation to assess the change in their quality of life as compared to baseline or prior to disease onset by using Aortic Disease Quality of Life (ADQoL) instrument and the validated general health related quality of life instrument called Short Form -12 (SF-12). The ADQoL is an instrument that measures the quality of life in 5 major domains - physical limitations, social limitations, general health perceptions, emotional limitations, and aortic-disease specific limitations. Lower scores on individual subscales and overall are deemed to be poor quality of life and higher scores indicate good quality of life. the SF-12 is also designed to assess general health related quality of life and is also scored and assessed similarly, i.e, higher scores indicate good general health related quality of life and measures health perception, physical, emotional, and social limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Kristofer M Charlton-Ouw, MD, FACS, Principal Investigator — University of Texas Health Science Center, UT Medical School Department of Cardiothoracic and Vascular Surgery, Houston
Locations (2):
- United States (2):
  - Department of Cardiothoracic and Vascular Surgery and Memorial Hermann Heart and Vascular Institute - Texas Medical Center, Houston, Texas
  - Department of Cardiothoracic and Vascular Surgery; Memorial Hermann Hospital Southeast, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be made available following IRB approval

REFERENCES:
- [Background] Afifi RO, Sandhu HK, Leake SS, Boutrous ML, Kumar V 3rd, Azizzadeh A, Charlton-Ouw KM, Saqib NU, Nguyen TC, Miller CC 3rd, Safi HJ, Estrera AL. Outcomes of Patients With Acute Type B (DeBakey III) Aortic Dissection: A 13-Year, Single-Center Experience. Circulation. 2015 Aug 25;132(8):748-54. doi: 10.1161/CIRCULATIONAHA.115.015302. PMID 26304666
- [Background] Nienaber CA, Rousseau H, Eggebrecht H, Kische S, Fattori R, Rehders TC, Kundt G, Scheinert D, Czerny M, Kleinfeldt T, Zipfel B, Labrousse L, Ince H; INSTEAD Trial. Randomized comparison of strategies for type B aortic dissection: the INvestigation of STEnt Grafts in Aortic Dissection (INSTEAD) trial. Circulation. 2009 Dec 22;120(25):2519-28. doi: 10.1161/CIRCULATIONAHA.109.886408. Epub 2009 Dec 7. PMID 19996018
- [Background] Nienaber CA, Kische S, Rousseau H, Eggebrecht H, Rehders TC, Kundt G, Glass A, Scheinert D, Czerny M, Kleinfeldt T, Zipfel B, Labrousse L, Fattori R, Ince H; INSTEAD-XL trial. Endovascular repair of type B aortic dissection: long-term results of the randomized investigation of stent grafts in aortic dissection trial. Circ Cardiovasc Interv. 2013 Aug;6(4):407-16. doi: 10.1161/CIRCINTERVENTIONS.113.000463. Epub 2013 Aug 6. PMID 23922146